CLINICAL TRIAL: NCT04748367
Title: Leveraging on Immersive Virtual Reality to Reduce Pain and Anxiety in Children During Immunization in Primary Care : A Pilot Randomised Control Trial
Brief Title: Leveraging on Immersive Virtual Reality to Reduce Pain and Anxiety in Children During Immunization in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SingHealth Polyclinics (Other)
Collaborators: Yoozoo Games Co., Ltd (Unknown); SingHealth DUKE-NUS Family Medicine Academic Clinical Programme (FM ACP) (Unknown)
Responsible Party: Principal Investigator, Chang Zi Ying, Principal Investigator, Deputy Clinic Director (SingHealth Polyclinic-Punggol branch), SingHealth Polyclinics
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019/2857
Record Dates: First submitted 2021-02-01; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Pain; Anxiety
Keywords: virtual reality; pain; anxiety; children; immunization
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Children wear VR headset during immunisation
  Interventions: Device: Virtual Reality Headset
- Control group (No Intervention): Children did not wear VR headset during immunisation( usual care)

INTERVENTIONS:
Device: Virtual Reality Headset — Virtual Reality Headset running SILVER software
  Arms: Intervention group

SUMMARY:
Paediatric immunization is often associated with significant fear and anxiety among children and their parents. Their distress can greatly affect their future adherence to the immunization schedule and the acceptance of recommended vaccines by physicians. This pilot was a single-centre, open label, randomised controlled trial to examine the use of VR analgesia in childhood immunization in primary care.The study primarily aimed to determine the feasibility of using immersive virtual reality (VR) during immunization in children by assessing the response rate of the participants during recruitment. The secondary outcome of the study was to determine the effectiveness of immersive VR in alleviating pain and anxiety among children during immunization compared to usual care without VR. It also aimed to determine the effectiveness of immersive VR in reducing anxiety among the parents and nurses during immunization procedure.

DETAILED DESCRIPTION:
This study primarily aimed to determine the feasibility of using immersive VR during immunization in children. The response rate of the recruitment was the feasibility assessment on whether children and parents were acceptable to the VR usage during immunization. The secondary outcome mainly focused on the clinical and safety outcomes of using immersive VR during immunization in preparation towards a larger randomized control trial. The secondary outcome of the study was the change in children's pain and anxiety scores using the Faces Pain Scale-Revised (FPS-R) and Children's Fear Scale (CFS) pre- and post-immunization. The other secondary outcome were the change in parent's and nurse's anxiety score using the Anxiety visual analogue scale (VAS).The nurses' acceptability, simplicity and willingness to use VR during immunization were also assessed in the study. Adverse events such as premature termination due to VR side effects in the children were also reported.

This pilot was a single-centre, open label, randomised controlled trial that was conceptualized as a proof of concept study to examine the use of VR analgesia in childhood immunization in primary care.

Study Setting and Population:

This study was conducted at a regional public primary care clinic (polyclinic) in Sengkang, which serves a population of about 240,000 inhabitants - of which children under the age of 9 years old account for 14.5% of them (second highest paediatric population in Singapore).The study populations included multi-ethnic Asian children aged 4 to 10 years, their parents and the registered nurses who administered their immunization at the polyclinic.

Sample Size:

Julious SA recommends a sample size of 12 per group as a rule of thumb for a pilot study. We recruited 30 children for this pilot study, with 15 in the intervention group (VR) and 15 in the control group to allow for estimated 3 children who may fail to use the VR during the immunization for whatever reasons.

Randomization:

Randomization was performed a-priori using a computer generated randomization system. The randomization sequences were concealed in a numbered, opaque envelope. Blinding of the subject was not possible in this study due to the nature of the intervention. After obtaining the consent and assent, the study team member retrieved the randomization envelopes to reveal the group assigned to the child.

Instrument to assess feasibility outcome:

The response rate of the recruitment of children and parents on this study was assessed.

Instruments to assess clinical outcome:

There are various self-reported measurement tools for pain assessment in children. We selected the FPS-R scale which is a validated and well-established psychometric test, recommended by various literature and International Association for the Study of Pain (IASP). FPS-R has strong positive correlations with the visual analogue scale (VAS) across the age of 4-16 years old.To date, there is no gold standard self-reported tools to measure children's anxiety during a needle procedure. We used the Children's Fear Scale (CFS) which was adapted from Faces Anxiety Scale that originally used in adult. Support was found for construct validity, test-retest reliability and inter-rater reliability for CFS during needle procedure among children. Anxiety VAS was used to assess anxiety in parents and nurses. The nurses' acceptability, simplicity and willingness to use VR during immunization were also assessed in the study, using a scale of 1 to 10.

VR equipment:

The VR equipment comprises an Oculus Quest headset (Facebook Technologies) which measures 8.7 x 7.6 x 4.1 inches and weighs 0.57kg. The field of angle is 100° with adjustable inter-pupil-distance (IPD) ranging from 58 to 72mm. The VR headset has an adjustable strap which can fit various head sizes.

VR software:

Evidence suggests that if the VR environment is individually tailored to user's age, gender, ethnicity, the VR analgesic effect will be enhanced. The VR software named SILVER (Soothing Immunization Leveraging on Virtual Reality Experience) was co-created by the two investigators with software engineers and virtual artist team from Yoozoo Games Co., Ltd in Singapore.

Recruitment procedure:

The clinical research coordinator (CRC) screened the appointment list of eligible children scheduled for their influenza or other childhood immunizations at the study site. When the child turned up for their immunization appointment, the CRC provided the parent or legal guardian with the study information and clarified their doubts before seeking their consent. They also spoke to the child on the potential use of the gadget used in the VR to seek their assent.

Written informed consent from the parent or legal guardian and assent from children were obtained prior to their study enrolment. The registered nurses involved also endorsed their consent to participate in the study. The study was conducted from September to December 2020.

Pre-intervention procedure:

The children in both groups rated their anticipatory pain score using the FPS-R scale and their anticipatory anxiety score using CFS. Their parents and respective attending nurses rated their anticipatory anxiety level using the Anxiety VAS before the immunization. The immunization room is cleared of any audio-visual equipment as a distraction in immunization.

Intervention group:

After revealing the allocation, the children allocated to the intervention group were briefed on the cartoon animation before they don the head-set. After the children entered the immunization room, the attending nurses completed their pre-procedure anxiety level using Anxiety VAS. The children donned the VR headset and viewed the VR animation. The animation can be viewed by the attending nurse via a tablet. At a specific juncture during the VR animation, the nurse administered the vaccine to the child. The duration of the storyline is about 2 minutes. At the end of each immunization, the VR headset will be cleaned and sanitized with standard infection control procedure in our institution.

Control group:

The children in control group underwent immunization as per usual care following our institution standard operating protocol. The nurse explained the immunization procedure to parents and children before the administration of the vaccine. The children in control group were not forbidden to use any distractions during immunization. Parents or additional nurses might be instructed to hold the child during the immunization procedure depending on the children's anxiety level to ensure accurate administration of the vaccine.

Statistical analysis:

All analyses were performed using IBM SPSS version 25.0. Both Intention to treat (ITT) and Per Protocol (PP) analysis were performed. Mann-Whitney U test was used to assess the difference in the change in anxiety and pain score in children, change in nurse's anxiety assessment and change in parent's anxiety assessment. Chi-square test and Fisher's exact test were used to assess the difference in the demographics of the two groups. Wilcoxon signed rank test was used to assess the difference in the nurses' experience of using the VR application. A p-value of less than 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Children of both gender and of any ethnicity are eligible to participate.
2. Parent (father or mother) or legal guardian or legal representative of the above children who accompany them to the polyclinic for immunization.
3. Registered nurses who are assigned to the immunization service stations during the period of the study.

Exclusion Criteria:

1. Children who are diagnosed with any disability or are deemed incapable of providing assent to the study will be excluded.
2. Children with pre-existing epilepsy/seizure or migraine
3. Caregivers including domestic helpers, grandparents, other relatives or nannies will be excluded.
4. Parent (father or mother) or legal guardian or legal representative who are affected by any disability which renders them incapable of providing consent will also be excluded.
5. Enrolled nurses or relief registered nurses at the study site will be excluded.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
Feasibility( the response rate of recruitment) using immersive VR during immunization in children, | within 10 minutes
  Response rate of recruitment (number of participants agree to participate divided by the total number of screened participants, expressed in % )

SECONDARY OUTCOMES:
Change children's pain score, using Faces Pain Scale-Revised (FPS-R) | 30 mins ( assess before and after immunisation)
  Faces Pain Scale-Revised (FPS-R) , in a scale of 0 to 10 (0 : no pain, 10: very much pain)
Change in children's anxiety score, using Children's Fear Scale (CFS) | 30 mins ( assess before and after immunisation)
  Children's Fear Scale (CFS) , in a scale of 0 to 4 (0: Not Scared at all , 4: Most Scared )
Change in parent's anxiety score, using Anxiety Visual Analogue Scale(VAS) | 30 mins ( assess before and after immunisation)
  Anxiety Visual Analogue Scale(VAS),in a scale of 0 to 10 ( 0: not anxious, 10: extremely anxious)
Change in nurses anxiety score, using Anxiety Visual Analogue Scale(VAS) | 30 mins ( assess before and after immunisation)
  Anxiety Visual Analogue Scale (VAS), in a scale of 0 to 10 ( 0: not anxious, 10: extremely anxious)
Simplicity of VR application during immunization by nurses | 5 mins
  Simplicity of VR application during immunization by nurses, in a scale of 1 to 10 ( 1: least simple, 10: most simple)
Acceptability to VR application during immunization by nurses | 5 mins
  Acceptability of VR application during immunization by nurses,in a scale of 1 to 10 ( 1: least acceptable, 10: most acceptable )
Willingness to use VR application in the future by nurses | 5 mins
  Willingness to use VR application in the future by nurses, in a scale of 1 to 10 (1: least willing, 10: most willing )

CONTACTS AND LOCATIONS:
Overall Officials: Zi Ying Chang, Principal Investigator — SingHealth Polyclinics
Locations (1):
- SingHealth Polyclinics-Sengkang, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang ZY, Kang GC, Koh EYL, Fong RJK, Tang J, Goh CK, Tan NC. Immersive Virtual Reality in Alleviating Pain and Anxiety in Children During Immunization in Primary Care: A Pilot Randomized Controlled Trial. Front Pediatr. 2022 Mar 25;10:847257. doi: 10.3389/fped.2022.847257. eCollection 2022. PMID 35402359